CLINICAL TRIAL: NCT02639767
Title: A Phase I Study of Concurrent Pemetrexed/Cisplatin With Pleural Intensity Modulated Radiation Therapy for Patients With Unresectable Malignant Pleural Mesothelioma
Brief Title: Concurrent Pemetrexed/Cisplatin With Pleural Intensity Modulated Radiation Therapy for Patients With Unresectable Malignant Pleural Mesothelioma
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-304
Record Dates: First submitted 2015-12-18; First posted 2015-12-24 (Estimated); Last update posted 2016-12-07 (Estimated); Status verified 2016-12

CONDITIONS: Malignant Pleural Mesothelioma
Keywords: Pemetrexed; Cisplatin; Intensity Modulated Radiation Therapy; 15-304
MeSH Terms: conditions — Mesothelioma, Malignant | interventions — Pemetrexed; Cisplatin

ARMS (1):
- pemetrexed/cisplatin with pleural IMRT (Experimental): This is a single institution phase I study of pemetrexed/cisplatin given concurrently with pleural intensity modulated radiation therapy (IMRT) in patients with unresectable malignant pleural mesothelioma (MPM). All patients will receive pleural intensity modulated radiation therapy (IMRT). Patients will be enrolled in cohorts of 3-6 at each dose level of pemetrexed/cisplatin, and dose escalation will proceed in a standard 3+3 fashion until the maximum tolerated dose (MTD) is identified.
  Interventions: Drug: Pemetrexed/Cisplatin; Radiation: Pleural Intensity Modulated Radiation Therapy; Device: MRI

INTERVENTIONS:
Drug: Pemetrexed/Cisplatin — Dose escalation of pemetrexed and cisplatin will follow the dose levels. The escalation will not exceed 500 mg/m^2 for pemetrexed in combination with 75 mg/m^2 of cisplatin even if the maximum tolerated dose is not identified. Each treatment cycle of chemotherapy will be 21 days. Patients will receive up to 2 cycles of chemotherapy during the radiation, and be followed for any DLT during the radiation therapy and for 12 weeks afterwards.
Radiation: Pleural Intensity Modulated Radiation Therapy — Pleura intensity modulated radiation therapy (IMRT) will be administered over approximately 6 weeks at 50.4 Gy in 28 fractions. The prescription radiation dose may anywhere between 45 and 50.4 Gy in 25 fractions if necessary to meet the normal tissue dose constraints.
Device: MRI — A pre-treatment MRI before chemo-RT will be acquired and will be used for target delineation. A three month post-treatment MRI will be acquired with the same protocol to assess the response from concurrent chemo-RT.

SUMMARY:
The purpose of this study is to evaluate the safety of combining chemotherapy at different doses with a specific type of radiation therapy delivered to the entire lining of the lung to find out what effects, if any, it has on people. This radiation technique is called pleural intensity modulated radiation therapy (IMRT). IMRT specifically targets the lining of the lung (pleura) where the cancer is and reduces the risk of damaging the lung itself. When given after chemotherapy, pleural IMRT has demonstrated promising results with respect to keeping mesothelioma under control longer. However, the investigators want to determine if giving pleural IMRT at the same time as chemotherapy is safe. If safe, further studies will be done to see if chemotherapy and pleural IMRT given at the same time keeps the tumor under control for a longer period of time than chemotherapy followed by pleural IMRT.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed diagnosis of malignant pleural mesothelioma at MSKCC
* No plans for surgical resection
* Stage T1-4, N0-3, M0
* No prior radiation therapy to the chest, breast or supraclavicular fossa that would limit radiation delivery to the full prescription dose
* Prior chemotherapy regimens ≤1
* Age ≥18 years
* Karnofsky performance status ≥ 80%
* Pulmonary function tests as follows: DLCO>50% predicted
* Adequate hematologic, hepatic, and renal function as indicated by the following laboratory values

  * Absolute neutrophil count ≥ 1,500/mcL
  * Platelets ≥ 100,000/mcL
  * Calculated creatinine clearance (CrCl) ≥ 45mL/min (using Cockcroft & Gault method)
  * Serum total bilirubin ≤ 1.5 x upper limit of normal (ULN) (unless known Gilbert's disease)
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x ULN

Exclusion Criteria:

* Pregnant or lactating women, or men or women not using effective contraception
* Patients with an active infection that requires systemic antibiotics, antiviral, or antifungal treatments
* Patients with a concurrent active malignancy (with the exception of skin cancer)
* Patients with serious unstable medical illness
* Patients with idiopathic pulmonary fibrosis
* Patients with NYHA heart failure class >2
* Patients with only one kidney that is ipsilateral to the mesothelioma
* Implanted pacemaker and/or defibrillator ipsilateral to the mesothelioma if it cannot be moved
* Patients meeting the following exclusion criteria will be excluded from the MRI portion only:
* Metallic implant, e.g. pacemaker, defibrillator
* Unmanageable claustrophobia
* High risk for nephrogenic systemic fibrosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-12; Primary Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicities (DLT) | up to 12 weeks
  The NCI Common Terminology Criteria for Adverse Events version 4.0 will be used to grade toxicities during the trial. DLTs are defined as any of the following events occurring during and for the first 12 weeks after completing pleural IMRT

CONTACTS AND LOCATIONS:
Overall Officials: Marjorie Zauderer, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (6):
- United States (6):
  - Memorial Sloan Kettering at Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Suffolk, Commack, New York
  - Memorial Sloan Kettering West Harrison, East White Plains, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Memoral Sloan Kettering Cancer Center at Phelps, Sleepy Hollow, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/